CLINICAL TRIAL: NCT06291701
Title: Investigation of the Relationship Between Scapular Endurance, Core Endurance, and Upper Extremity Functional Performance in Adolescent Tennis Players
Brief Title: The Relationship Between Scapular Endurance, Core Endurance, and Functional Performance in Adolescent Tennis Players
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Elif AYGUN POLAT, PhD, PT, Ordu University
Other Study IDs: ODUSBFFTR-ELIFAYGUNPOLAT-002
Record Dates: First submitted 2024-02-07; First posted 2024-03-04 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Athletic Injuries; Sports Physical Therapy
Keywords: core endurance; scapular endurance; adolescent tennis player; upper extremity functional performance
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Other: adolescent tennis player
  Interventions: Diagnostic Test: Assessment of scapular endurance; Diagnostic Test: Prone Bridge Test; Diagnostic Test: Side Bridge Test; Diagnostic Test: Closed Kinetic Chain Upper Extremity Stability Test; Diagnostic Test: Seated Medicine Ball Throw Test

INTERVENTIONS:
Diagnostic Test: Assessment of scapular endurance — For the assessment of scapular endurance, participants will be instructed to bend their arms and elbows while keeping a wooden rod placed between their elbows, pull a spring dynamometer placed between thei
Diagnostic Test: Prone Bridge Test — For the "Prone Bridge Test," participants will be instructed to lie face down with their hands and feet shoulder-width apart and then raise their bodies off the ground by lifting themselves up on their hands, forearms, and toes. A stopwa
Diagnostic Test: Side Bridge Test — For the "Side Bridge Test," participants will be asked to lie on their right side, supporting themselves on their forearm and elbow, and lift themselves off the ground. A stopwatch will be started, and the test will be terminated if there is any deviation from the position. The elapsed time will be recorded in seconds. The test will then be repeated on the left side.
Diagnostic Test: Closed Kinetic Chain Upper Extremity Stability Test — For the Closed Kinetic Chain Upper Extremity Stability Test, participants will be asked to assume a push-up position on a flat surface with their hands placed on two parallel lines drawn 90 cm apart. They will then be instructed to touch one hand to the other hand's side as many times as possible within 15 seconds. The test will be repeated three times, and the average of the scores will be calculated.
Diagnostic Test: Seated Medicine Ball Throw Test — For the "Seated Medicine Ball Throw Test," participants will be asked to sit on the ground with their back, shoulders, and head against the wall. Holding a 2 kg medicine ball with both hands, they will start with their elbows bent and arms at their sides, then extend their elbows to throw the ball forward as far as possible. The distance between the wall and the point where the ball lands will be recorded. The test will be performed three times, and the average will be calculated.

SUMMARY:
This study aims to examine the relationship between scapular endurance, core endurance, and upper extremity performance in adolescent tennis players. The hypothesis of this study is that better scapular/core endurance in adolescent tennis players is associated with better upper extremity performance. Establishing this relationship will contribute to identifying the exercise training necessary to improve upper extremity performance in tennis players.

DETAILED DESCRIPTION:
Tennis is a sport characterized by coordinated, repetitive, and powerful movements along the kinetic chain. Being both overhead and rotational, achieving a good shot in tennis involves transferring high forces and energy from the lower extremities to the upper extremities through the trunk. In this context, core muscles play a crucial role in athletic performance by stabilizing the shoulder girdle, pelvis, and spine, acting as a pivot point for extremity movements. Therefore, good core strength is essential during a stroke. Additionally, as the acceleration of the ball is influenced by both maximum external and internal rotation of the shoulder, tennis players require good shoulder mobility and stability. In this regard, the scapula in the shoulder girdle provides a stable foundation for the glenohumeral mobility necessary for the shot. Both the core and scapular regions serve as pivot points for upper extremity functional activities. Therefore, this study aims to examine the relationship between scapular endurance, core endurance, and upper extremity performance in adolescent tennis players. The hypothesis of this study is that better scapular/core endurance in adolescent tennis players is associated with better upper extremity performance. Establishing this relationship will contribute to identifying the exercise training necessary to improve upper extremity performance in tennis players.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent tennis players

Exclusion Criteria:

* Athletes with a history of musculoskeletal injury or surgery in the last year that would prevent the tests from being performed
* Athletes who feel pain in the trunk and lower extremities during the tests

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescent tennis players
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Prone Bridge Test | first day, in an average of one hour
  For the measurement of core endurance, Prone Bridge Test will be applied.For the "Prone Bridge Test," participants will be instructed to lie face down with their hands and feet shoulder-width apart and then raise their bodies off the ground by lifting themselves up on their hands, forearms, and toes. A stopwatch is started, and the test is terminated if there is any deviation from the proper position. The elapsed time is recorded in seconds.
Side Bridge Test | first day, in an average of one hour
  For the measurement of core endurance, Side Bridge Test will be applied. For the "Side Bridge Test," participants will be asked to lie on their right side, supporting themselves on their forearm and elbow, and lift themselves off the ground. A stopwatch will be started, and the test will be terminated if there is any deviation from the position. The elapsed time will be recorded in seconds. The test will then be repeated on the left side.
Scapular Endurance Values | first day, in an average of one hour
  For the assessment of scapular endurance, participants will be instructed to bend their arms and elbows while keeping a wooden rod placed between their elbows, pull a spring dynamometer placed between their hands without dropping the wooden rod, and maintain this position. A stopwatch will be started, and the elapsed time will be recorded in seconds.
Closed Kinetic Chain Upper Extremity Stability Test | first day, in an average of one hour
  For the Closed Kinetic Chain Upper Extremity Stability Test, participants will be asked to assume a push-up position on a flat surface with their hands placed on two parallel lines drawn 90 cm apart. They will then be instructed to touch one hand to the other hand's side as many times as possible within 15 seconds. The test will be repeated three times, and the average of the scores will be calculated.
Seated Medicine Ball Throw Test | first day, in an average of one hour
  For the "Seated Medicine Ball Throw Test," participants will be asked to sit on the ground with their back, shoulders, and head against the wall. Holding a 2 kg medicine ball with both hands, they will start with their elbows bent and arms at their sides, then extend their elbows to throw the ball forward as far as possible. The distance between the wall and the point where the ball lands will be recorded. The test will be performed three times, and the average will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Sevim Beyza OLMEZ, PhD, Principal Investigator — Karamanoğlu Mehmetbey University; Zeynep Hazar, Prof, Study Director — Gazi University
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.